CLINICAL TRIAL: NCT05014958
Title: The Effect of 6-week Whole Body Vibration Training on Trunk Muscle Strength, Body Composition and Performance Parameters
Brief Title: The Effect of Whole Body Vibration Training on Trunk Muscle Strength, Body Composition and Performance Parameters
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Ali ZORLULAR, Principal Investigator, Physiotherapist, Gazi University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2020-438
Record Dates: First submitted 2021-08-04; First posted 2021-08-20 (Actual); Last update posted 2023-12-05 (Actual); Status verified 2023-12

CONDITIONS: Health, Subjective

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 40 hz frequency exercise group (Experimental): Individuals in this study group will receive exercise training at 40 hz frequency on whole body vibration device.
  Interventions: Other: Exercise training on whole body vibration
- 25 hz frequency exercise group (Experimental): Individuals in this study group will receive exercise training at 25 hz frequency on whole body vibration device.
  Interventions: Other: Exercise training on whole body vibration
- 0 hz frequency exercise group (Active Comparator): Individuals in this study group will receive exercise training at 0 hz frequency on whole body vibration device.
  Interventions: Other: Exercise training on whole body vibration

INTERVENTIONS:
Other: Exercise training on whole body vibration — Participants will be included in the 6-week exercise training on whole body vibration

SUMMARY:
Whole body vibration (WBV) trainings are widely used in the field of sports medicine and rehabilitation. It is accepted that these trainings are a modality that can safely increase muscular activation and performance. However, although many exercise models have been tried on vibration platforms, a standard WBV program for trunk muscles has not been established. A total of 45 healthy individuals will be included in the study. Participants will be divided into 3 groups. Group 1 will perform exercises at 40hz frequency, group 2 will perform exercises at 25hz frequency on WBV. The control group will perform the same exercises at 0 Hz. The training will last 6 weeks and each session consists of 5 exercises.The training consists of basic core exercises that the individual does with his or her own body weight. Each training session is approximately 30 minutes. All participants will be evaluated using an isokinetic strength test with a Cybex dynamometer at the beginning and at the end of the additional treatment protocol. In addition, balance, body composition and anaerobic performance of individuals will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults
* The age range should be between 20-35

Exclusion Criteria:

* Having an orthopedic problem
* Having orthopedic surgery in the last 6 months
* Doing daily exercise and sport

Ages: 20 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2021-05-17 (Actual); Primary Completion 2021-12-17 (Actual); Study Completion 2021-12-30 (Actual)

PRIMARY OUTCOMES:
Muscle Strength Assesment | 20 Minutes
  Muscle Strength Assesment will be evaluated using isokinetic dynamometer

SECONDARY OUTCOMES:
Balance Assesment | 12 Minutes
  Posturography will be used to assess static balance
Body Composition Assesment | 3 Minutes
  Body Composition will be evaluated using bioelectrical impedance analyzer
Anaerobic Power Assesment | 5 Minutes
  Anaerobic Power will be evaluated using 3D accelerometer

CONTACTS AND LOCATIONS:
Overall Officials: Ali Zorlular, Msc, Principal Investigator — Gazi University
Locations (1):
- Gazi University, Ankara, Turkey (Türkiye)

REFERENCES:
- [Derived] Zorlular A, Kafa N, Guzel NA. Effects of 6-Week Whole-Body Vibration Training on Isokinetic Trunk Muscle Strength, Postural Stability, and Jump Performance in Female Adults - A Randomized Controlled Trial. Res Q Exerc Sport. 2025 Sep;96(3):523-531. doi: 10.1080/02701367.2024.2447502. Epub 2025 Jan 31. PMID 39889143